CLINICAL TRIAL: NCT06700187
Title: Effects of Sitting Interruption Frequency on Cognitive Function and Glucose Metabolism: A Randomized, Controlled Cross-over Study Involving Young Sedentary Adults
Brief Title: Frequency of Interrupting Sitting and Cognitive Function
Acronym: FISCF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: NL86254.068.24; CCMO, WMO (Registry Identifier: NL-OMON57014)
Record Dates: First submitted 2024-11-12; First posted 2024-11-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Sedentary Behaviors; Breaking Prolonged Sitting With Physical Activity
Keywords: Sedentary behavior; sitting interruptions; cognition; glucose metabolism
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interrupting sitting (Experimental): Participants will engage in low-intensity walking breaks in different frequencies for 4.5 hours
  Interventions: Other: Interrupting sitting with walking breaks
- Control (No Intervention): Paticipants will remain seated for 4.5 hours

INTERVENTIONS:
Other: Interrupting sitting with walking breaks — Participants will engage in 27 minutes walking in different frequencies, including short breaks (walk 1 minute every 10 minutes), moderate breaks (walk 3 minutes every 30 minutes), and long breaks (walk 27 minutes in one time during the intervention).
  Arms: Interrupting sitting

SUMMARY:
Rationale: Sedentary behavior (SB) has been associated with impaired cognitive function in elderly, and negatively impacts glucose metabolism. Interrupting sitting with physical activity (PA) bouts may exert beneficial effects on cognitive function via an improved glucose metabolism. Nevertheless, the impact of breaking up prolonged sitting with various frequencies of PA bouts remains unexplored in young sedentary adults. Moreover, we hypothesize that the pattern of the breaks modifies the effects. Thus, randomized controlled trials (RCTs) are highly needed to investigate the effects of interrupting sitting with different frequencies of PA on cognitive function and glucose metabolism. We now hypothesize that interrupting sitting with different frequencies of walking breaks differentially affects cognitive function and glucose metabolism.

Objective: The aim is to investigate the effects of breaking up sitting with different frequencies of PA bouts on cognitive function and glucose metabolism in young sedentary adults.

Study design: A randomised, controlled cross-over study will be performed, consisting of four interventions in a counterbalanced order: uninterrupted prolonged sitting, short breaks, moderate breaks, and long breaks.

Intervention: Participants will complete four conditions in a randomized, counterbalanced order: sitting (uninterrupted prolonged sitting without any interruptions), short breaks (walk 1 minute every 10 minutes), moderate breaks (walk 3 minutes every 30 minutes), and long breaks (walk 27 minutes during the intervention). Each condition lasts 4.5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-35 years;
* BMI between 18.5-24.9 kg/m2;
* SB, i.e. sitting for an average of at least 9 hours per day;
* Physically inactive, i.e. engaging in exercise for less than 2 to 3 times per week;
* Stable body weight (weight gain or loss < 3 kg in the past three months);
* Willingness to engage in four 6-hour laboratory visits;
* No difficult cannulation.

Exclusion Criteria:

* Not sedentary, i.e. sitting for less than an average of 9 hours per day;
* Physically active, i.e. engaging in exercise for more than 3 times a week;
* Abuse of drugs;
* Use medication to treat BP, lipid, or glucose metabolism;
* Pregnant females.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Mental flexibility | baseline and 5 hours post baseline
  It will be assessed using the computer-based Trial Making Test

SECONDARY OUTCOMES:
Interference | baseline and 5 hours post baseline
  Interference is assessed by the computer-based Stroop task
Memory | baseline and 5 hours post baseline
  Memory is assessed by the computer-based n-Back Test
Attention | baseline and 5 hours post baseline
  Attention is assessed by the paper-based d2 attention Test
Glucose metabolism | baseline, 30 minutes, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, and 5 hour post baseline
  Concentration of plasma glucose will be tested.
Glucose metabolism | baseline, 30 minutes, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, and 5 hour post baseline
  Concentration of serum insulin will be tested.
Serum brain-derived neurotrophic factor (BDNF) | baseline, 2 hour, 3 hour, and 5 hour post baseline
  Concentration of serum BDNF, as one of the exploratory outcomes will be tested.
Blood lipids | baseline, and 5 hours post baseline
  As exploratory outcomes, concentration of serum total cholesterol (TC), and high-density lipoprotein cholesterol (HDL-C) will be tested.
Serum triacylglycerol (TAG) | baseline, 30 minutes, 1 hour, 1.5 hour, 2 hour, 3 hour, 4 hour, and 5 hour post baseline
  As another exploratory outcome, concentration of serum TAG will be tested.
Mood | baseline and 5 hours post baseline
  Short version of Profile of Mood States (POMS) questionnaire will be used to test mood.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition and movement science, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individuals wanting access to IPD should contact the principal investigator (hans.savelberg@maastrichtuniversity.nl)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting after 6 months of publication
Access Criteria: Available to all researchers interested in interrupting sitting studies

REFERENCES:
- [Background] Wheeler MJ, Green DJ, Cerin E, Ellis KA, Heinonen I, Lewis J, Naylor LH, Cohen N, Larsen R, Dempsey PC, Kingwell BA, Owen N, Dunstan DW. Combined effects of continuous exercise and intermittent active interruptions to prolonged sitting on postprandial glucose, insulin, and triglycerides in adults with obesity: a randomized crossover trial. Int J Behav Nutr Phys Act. 2020 Dec 14;17(1):152. doi: 10.1186/s12966-020-01057-9. PMID 33308235
- [Background] Homer AR, Taylor FC, Dempsey PC, Wheeler MJ, Sethi P, Townsend MK, Grace MS, Green DJ, Cohen ND, Larsen RN, Kingwell BA, Owen N, Dunstan DW. Frequency of Interruptions to Sitting Time: Benefits for Postprandial Metabolism in Type 2 Diabetes. Diabetes Care. 2021 Jun;44(6):1254-1263. doi: 10.2337/dc20-1410. Epub 2021 Apr 26. PMID 33905343
- [Background] Duran AT, Friel CP, Serafini MA, Ensari I, Cheung YK, Diaz KM. Breaking Up Prolonged Sitting to Improve Cardiometabolic Risk: Dose-Response Analysis of a Randomized Crossover Trial. Med Sci Sports Exerc. 2023 May 1;55(5):847-855. doi: 10.1249/MSS.0000000000003109. Epub 2023 Jan 12. PMID 36728338
- [Background] Wheeler MJ, Green DJ, Ellis KA, Cerin E, Heinonen I, Naylor LH, Larsen R, Wennberg P, Boraxbekk CJ, Lewis J, Eikelis N, Lautenschlager NT, Kingwell BA, Lambert G, Owen N, Dunstan DW. Distinct effects of acute exercise and breaks in sitting on working memory and executive function in older adults: a three-arm, randomised cross-over trial to evaluate the effects of exercise with and without breaks in sitting on cognition. Br J Sports Med. 2020 Jul;54(13):776-781. doi: 10.1136/bjsports-2018-100168. Epub 2019 Apr 29. PMID 31036563
- [Background] Wu Y, Van Gerven PWM, de Groot RHM, Eijnde BO, Winkens B, Savelberg HHCM. Effects of breaking up sitting with light-intensity physical activity on cognition and mood in university students. Scand J Med Sci Sports. 2023 Mar;33(3):257-266. doi: 10.1111/sms.14277. Epub 2022 Dec 1. PMID 36434768